CLINICAL TRIAL: NCT03274323
Title: Trabeculectomy Versus 2-iStent and Prostaglandin Study
Acronym: TIPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty obtaining IDE by the FDA. Currently not worthwhile to pursue further.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00146334
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 2 iStent with travoprost or latanoprost (Experimental): 2 iStents will be injected into the trabecular meshwork and patients will be administered topical latanoprost or travoprost following surgery
  Interventions: Device: iStent and travoprost or latanoprost
- trabeculectomy (Active Comparator): Standard trabeculectomy
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Device: iStent and travoprost or latanoprost — 2 iStents will be inserted and patients will be started on travoprost or latanoprost following the procedure
  Arms: 2 iStent with travoprost or latanoprost
Procedure: Trabeculectomy — Standard trabeculectomy
  Arms: trabeculectomy

SUMMARY:
Investigators hypothesize that the synergistic action of iStent in increasing aqueous outflow through the trabecular meshwork and use of prostaglandin analog such as travoprost or latanoprost to increase uveoscleral outflow will achieve good Intra-ocular Pressure (IOP) control with minimal complications in Primary Open Angle Glaucoma (POAG) patients with suboptimal IOP on 2 or more medications compared to mitomycin C (MMC) augmented trabeculectomy.

DETAILED DESCRIPTION:
This will be a prospective randomized controlled study.

20 phakic or pseudophakic open angle glaucoma patients with an IOP in the range of 18-30 mmHg on 2 or more topical glaucoma medications will be randomly selected to undergo either (1) mitomycin-augmented trabeculectomy or (2) placement of 2 iStent devices and initiation of a daily prostaglandin analog. This study is looking at the combined effects of the 2 iStents and a prostaglandin analog as a method to achieve low IOP. At 3 months (+/- 2 weeks) postoperatively, the iStent patients will be left only on the prostaglandin analog with a washout performed for any other hypotensive medication used. Patients who had a trabeculectomy will be have a terminal washout of all IOP-lowering medications at 3 months (+/- 2 weeks) post-surgery. The IOP will then be measured for both groups at 4 months (+/- 3 weeks) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have mental capacity to give consent
* Age >= 21 years
* Pseudophakic or phakic without visually significant cataract
* Open angle glaucoma
* IOP in the range of 18-30 mmHg with 2 or more topical medications
* Cup-disc ratio =< 0.9
* Best corrected visual acuity of 20/100 or better

Exclusion Criteria:

* Inability to give consent
* Inability to tolerate or presence of allergy to prostaglandin analogs
* Patient preference for non-surgical treatment or preference for either of the recommended surgical modalities in the study
* Age < 21 years
* Visually significant cataract that would benefit from cataract surgery, as determined by the treating surgeon in consultation with the patient
* Secondary glaucoma or angle closure glaucoma
* Aphakia
* Prior glaucoma incisional surgery (trabeculectomy, tube surgery, other Microinvasive Glaucoma Surgery (MIGS) surgeries, deep sclerectomy)
* Prior laser trabeculoplasty < 90 days prior to screening or absolute failure of prior laser trabeculoplasty.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
IOP <= 18 mmHg | Post surgery month 4
  IOP
IOP <= 15 mmHg | Post surgery month 4
  IOP
IOP >= 20% reduction from untreated baseline | Post surgery month 4
  IOP

IPD SHARING:
Plan to Share IPD: No